CLINICAL TRIAL: NCT00772395
Title: Can Risedronate Prevent Periprosthetic Bone Loss After Total Hip Arthroplasty. A Randomized, Double-blind, Placebo-controlled, Parallel-group Study
Brief Title: Can Risedronate Prevent Periprosthetic Bone Loss After Total Hip Arthroplasty
Acronym: PREVENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Danderyd Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Olof Skoldenberg, Consulatant Orthopaedic Surgeon, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-745/4; 04-745/4
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Bone Loss
Keywords: Periprosthetic bone loss risedronate bisphosphonates
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risedronate (Active Comparator)
  Interventions: Drug: Risedronate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Risedronate — 35 mg given once weekly start on 2nd postoperative day for 26 weeks (6 months)
  Arms: Risedronate
Drug: Placebo — Placebo given once weekly start on 2nd postoperative day for 26 weeks (6 months)
  Arms: Placebo

SUMMARY:
Can risedronate given once weekly for 6 months prevent periprosthetic bone loss after uncemented total hip arthroplasty?

DETAILED DESCRIPTION:
Periprosthetic bone loss after total hip arthroplasty is the main factor in limiting the longevity of implants used for treatment of osteoarthritis. Bone loss leads to implant destabilization. Bisphosphonates, given for approximately 6 months after THA man prevent this bone loss and lead to longer implant fixation and lower incidence of aseptic prosthesis loosening. We perform a clinical trial with risedronate to investigate if we can influence periprosthetic bone loss around a uncemented femoral stem.

ELIGIBILITY:
Inclusion Criteria:

* Patients on the waiting list for a total hip arthroplasty
* Primary osteoarthritis
* Osteoarthritis secondary to congenital dislocation of the hip

Exclusion Criteria:

* Rheumatoid arthritis
* Bisphosphonate treatment
* Osteomalacia
* Hypocalcemia
* Previous surgery of the affected hip

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2006-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Can risedronate given once weekly for 6 months prevent periprosthetic bone loss up to 2 years after uncemented total hip arthroplasty | 4 years

SECONDARY OUTCOMES:
Can risedronate reduce migration of a uncemented femoral stem | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Olof G Sköldenberg, MD, Principal Investigator — Department of clinical sciences at Danderyd hospital
Locations (1):
- Orthopaedic department, Danderyd Hospital, Stockholm, Stockholm County, Sweden